CLINICAL TRIAL: NCT01437046
Title: Doxazosin an a1 Antagonist for Alcohol Dependence
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Carolina L Haass-Koffler, PI, Brown University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1101000328; 1R21AA019994-01A1 (NIH)
Record Dates: First submitted 2011-09-19; First posted 2011-09-20 (Estimated); Last update posted 2025-08-18 (Actual); Status verified 2016-02

CONDITIONS: Alcohol Dependence; Anxiety
Keywords: Alcohol drinking; Alcohol craving
MeSH Terms: conditions — Alcoholism; Anxiety Disorders; Alcohol Drinking | interventions — Doxazosin; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (2):
- Doxazosin (Experimental): Doxazosin Capsule 16mg/day 10 weeks.
  Interventions: Drug: Doxazosin
- Placebo (Placebo Comparator): Placebo (lactose capsules designed to be the same as experimental drug given the same exact way over 10 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Doxazosin — Doxazosin were prepared as opaque capsules by a compounding pharmacy and inserted into blister packs. Consistent with the recommended titration, doxazosin was titrated up to 16 mg daily (or maximum tolerable dose) during the first 4 weeks. A 1-week downward titration for safety reasons was also planned. Study medication adherence was assessed by self-report and pill count. Additionally, capsules contained 25mg riboflavin as a marker of adherence through urine sample.
  Other Names: Cardura
  Arms: Doxazosin
Drug: Placebo — Matched placebo were prepared as opaque capsules by a compounding pharmacy and inserted into blister packs. Consistent with the recommended titration, doxazosin or matched placebo was titrated up to 16 mg daily (or maximum tolerable dose) during the first 4 weeks. A 1-week downward titration for safety reasons was also planned. Study medication adherence was assessed by self-report and pill count. Additionally, capsules contained 25mg riboflavin as a marker of adherence through urine sample.
  Other Names: Lactose
  Arms: Placebo

SUMMARY:
Norepinephrine system represents an important treatment target for alcohol dependence (AD) and the α1 -blocker prazosin may reduce alcohol drinking in rodents and alcoholic patients. The α1 -blocker doxazosin demonstrates a more favorable pharmacokinetic profile than prazosin, but has never been studied for AD. A double-blind placebo-controlled randomized clinical trial was designed in AD individuals seeking outpatient treatment. Doxazosin or matched placebo was titrated to 16 mg/day (or maximum tolerable dose). Drinks per week (DPW) and heavy drinking days (HDD) per week were the primary outcomes. Family history density of alcoholism (FHDA), severity of AD and gender were a priori moderators.

DETAILED DESCRIPTION:
Pre-clinical and clinical evidence has clearly demonstrated that the noradrenergic (NE) system is involved in the neurobiology of AD, thus representing an interesting new pharmacotherapy target and the theoretical rationale for this proposal. Consistent with the concept that the NE system may represent a new pharmacological target for AD, recent studies have shown that the prototype alpha-1 NE receptor antagonist prazosin reduces alcohol drinking in different animal models. Furthermore, clinical evidence has also confirmed that prazosin appears to be efficacious in reducing alcohol consumption in alcohol-dependent individuals. While prazosin has a significant side effect profile and must be taken three times a day, no other α1-blockers have been investigated in alcohol research. Prazosin is a short-acting α1-blocker approved to treat hypertension (HTN) and benign prostatic hyperplasia (BPH). After the approval of prazosin in the 70's, other selective α1-blockers have been developed to treat HTN and/or BPH. Among them, doxazosin has shown a more manageable and safer profile than prazosin. In fact, doxazosin is a long-acting α1-blocker, thus it is taken only once/day. Doxazosin is also less likely to give hypotensive side-effects. Thus, doxazosin is more commonly used in clinical practice to treat HTN and/or BPH, than short-acting α1-blockers, such as prazosin. Poor adherence to medications and/or side-effects represent important factors limiting the effectiveness of pharmacotherapies for patients with AD. If effective for AD, doxazosin may represent a simple, manageable and safe medication, which might be more easily transferable to clinical practice. However, doxazosin has never been tested in AD. This project is a 10-week, double-blind, placebo-controlled, between-subject randomized clinical trial with doxazosin (16mg once/day) in alcohol dependent (AD) individuals. This study attempts to address whether doxazosin is an effective and safe pharmacotherapy for AD.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18
* females must be post-menopausal for ≥1 year, surgically sterile, or practicing a birth control before entry and throughout the study; have a negative urine pregnancy test at screening and before randomization
* good health (confirmed by medical history, physical, ECG, blood/urine labs)
* DSM-IV diagnosis of AD
* average of ≥4 drinks/d for women and ≥5 drinks/d for men during 30 days within the 90 days prior to screening
* desire to reduce or quit drinking.

Exclusion Criteria:

* females who are of child bearing potential and not practicing effective birth control
* lifetime DSM-IV diagnosis of schizophrenia, bipolar disorder, or other psychosis
* recent (past 6 months) DSM-IV diagnosis of any anxiety disorder or major depression
* in the investigators' opinion, risk of suicide (e.g. active plan, or recent attempt in last year)
* DSM-IV diagnosis of dependence on any psychoactive substance other than alcohol and nicotine
* positive urine screen for any illegal substance other than marijuana
* history of hospitalization for alcohol intoxication delirium, seizure or alcohol withdrawal delirium
* Clinical Institute Withdrawal Assessment for Alcohol (CIWA-Ar) score ≥10, at any assessment
* treatment with naltrexone, acamprosate, topiramate, disulfiram within 1 month prior to Wk 00
* current use of psychotropic medications or drugs that interfere with doxazosin's metabolism
* use of PDE5 inhibitor erectile dysfunction drugs (e.g. sildenafil)
* treatment with any antihypertensive drug and/or any α-blocker for BPH or sleep problems (e.g. trazodone)
* baseline hypotension
* history of allergy to any α-blocker
* contraindications to take doxazosin (history of fainting and/or syncopal attacks, heart failure, significant liver diseases)
* serious illnesses, e.g. kidney failure, epilepsy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-11-01 (Actual); Primary Completion 2013-08-01 (Actual); Study Completion 2015-03-01 (Actual)

PRIMARY OUTCOMES:
drinking days per week (DDW) | 16 weeks
  whether doxazosin, as compared to placebo, decreases the number of drinking days per week (DDW), as measured by the timeline follow-back (TLFB). A drink is defined as a Standard Drinking Unit (SDU).
drinks per week (DPW) | 16 weeks
  whether doxazosin, as compared to placebo, decreases the number of drinks per week (DPW), measured by the TLFB

SECONDARY OUTCOMES:
alcohol craving | 16 weeks
  whether doxazosin, as compared to placebo, results in diminished alcohol craving, as measured by the Obsessive Compulsive Drinking Scale (OCDS)
anxiety | 16 weeks
  whether doxazosin, as compared to placebo, results in diminished anxiety scores, measured by the Hamilton Anxiety Scale (HAMA).
Adverse Events | 16 weeks
  whether doxazosin, as compared to placebo, increases the frequency and intensity of Adverse Events (AE).

CONTACTS AND LOCATIONS:
Overall Officials: GEORGE A KENNA, PhD RPh, Principal Investigator — Brown University
Locations (1):
- Brown University Center for Alcohol and Addiction Studies, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
email the PI to make arrangements for sharing the available database.

REFERENCES:
- [Background] Kenna GA, Haass-Koffler CL, Zywiak WH, Edwards SM, Brickley MB, Swift RM, Leggio L. Role of the alpha1 blocker doxazosin in alcoholism: a proof-of-concept randomized controlled trial. Addict Biol. 2016 Jul;21(4):904-14. doi: 10.1111/adb.12275. Epub 2015 Jun 2. PMID 26037245